CLINICAL TRIAL: NCT06957964
Title: Prophylactic Negative Pressure Wound Therapy in Laparotomy Wounds: A Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Hamail Khanum (Other)
Responsible Party: Sponsor-Investigator, Dr Hamail Khanum, Head of Department Surgery, Gulab Devi Hospital
Organization: Gulab Devi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 280
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Wound; Infection Prevention; Negative Pressure Wound Therapy
MeSH Terms: conditions — Wounds and Injuries | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with Negative Pressure Wound Therapy (Experimental): In group A, Negative Pressure Wound Therapy will be applied at end of laparotomy. Participants will be shifted to post-surgical wad for 72 hours and then will be discharged with prescription of standard antibiotics course. Patients will be followed-up in OPD for 30 days and will be assessed in terms of surgical site infection and re operation.
  Interventions: Other: Negative Pressure Wound Therapy; Drug: Standard Antibiotic Treatment
- Participants without Negative Pressure Wound Therapy (Experimental): In group B, Negative Pressure Wound Therapy will be applied at end of laparotomy. Participants will be shifted to post-surgical wad for 72 hours and then will be discharged with prescription of standard antibiotics course. Patients will be followed-up in OPD for 30 days and will be assessed in terms of surgical site infection and re operation.
  Interventions: Drug: Standard Antibiotic Treatment

INTERVENTIONS:
Other: Negative Pressure Wound Therapy — Negative Pressure Wound Therapy is an intervention in which a suction is applied at applied thus creating a negative pressure which not only removes any exudate but also aids in formation of granulation tissue. NPWT is provided along with empirical prophylactic antibiotics
  Arms: Participants with Negative Pressure Wound Therapy
Drug: Standard Antibiotic Treatment — According to hospital antibiogram, empirical antibiotics are given prophylactically

SUMMARY:
Total 70 participants meeting selection criteria will be enrolled in the study from operational theatre. They will be randomly divided in two groups by using lottery method. In group A, Negative Pressure Wound Therapy will be applied at end of procedure. In group B, no Negative Pressure Wound Therapy will be placed. They will be shifted to post-surgical wad for 72 hours and then will be discharged with prescription of standard antibiotics and will be followed-up in OPD for 30 days. If patient will develop surgical site wound infection, then it will be noted. If infection will not be cured with antibiotics course, then re-operation will be done. Patients complications will be managed as per hospital protocol. All this information will be recorded in proforma.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age between 20 to 70 years, both genders
* Undergoing laparotomy under general anaesthesia
* ASA I-II

Exclusion Criteria:

* Patients who did not complete the follow up instructions
* Pregnant patients
* Patients already undergone a relook laparotomy, if their abdomen is left open or if unable to adhere

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | 03 Months
  It will be labelled if there will be presence of pus and pus discharge from wound site, confirmation of presence of pathogen through culture along with presence of pain, swelling, tenderness at wound site on physical examination during 15-30 days of surgery.

SECONDARY OUTCOMES:
Re Operation | 03 Months
  It will be labelled if patient will undergo surgery due to severe surgical site wound infection that develop during 15-30 days of surgery and not healed with antibiotics course.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Dr Maratab Ali, MBBS FCPS, Study Director — Gulab Devi Hospital
Locations (1):
- Gulab Devi Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No